CLINICAL TRIAL: NCT02222155
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Assessment Phase 2 Study to Evaluate the Safety and Efficacy of CCX168 in Subjects With Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of CCX168 in ANCA-Associated Vasculitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL003_168; #FD-R-5414 (Other: Orphan Products Development Grant)
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: ANCA-associated Vasculitis
Keywords: ANCA-associated vasculitis; complement; vasculitis; C5aR
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — avacopan; Rituximab; Glucocorticoids; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CCX168 low dose plus standard of care (Active Comparator): Capsule, 10 mg, twice daily + standard of care for 12 weeks
  Interventions: Drug: CCX168 10 mg, twice daily, plus cyclophosphamide/rituximab plus glucocorticoids
- CCX168 high dose plus standard of care (Active Comparator): Capsule, 30 mg, twice daily + standard of care for 12 weeks
  Interventions: Drug: CCX168 30 mg, twice daily, cyclophosphamide/rituximab plus glucocorticoids
- Placebo, twice daily + standard of care (Placebo Comparator): Capsule, placebo, twice daily + standard of care for 12 weeks
  Interventions: Other: Placebo, twice daily, plus cyclophosphamide/rituximab plus glucocorticoids

INTERVENTIONS:
Drug: CCX168 10 mg, twice daily, plus cyclophosphamide/rituximab plus glucocorticoids
  Arms: CCX168 low dose plus standard of care
Drug: CCX168 30 mg, twice daily, cyclophosphamide/rituximab plus glucocorticoids
  Arms: CCX168 high dose plus standard of care
Other: Placebo, twice daily, plus cyclophosphamide/rituximab plus glucocorticoids
  Arms: Placebo, twice daily + standard of care

SUMMARY:
The aim of this trial is to test the safety and efficacy of two dose regimens of the complement C5a receptor CCX168 in patients with anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV).

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Complement 5a and its receptor C5aR (CD88) is involved in the pathogenesis of anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis. This is a randomized, double-blind, placebo-controlled Phase 2 study to evaluate the safety and efficacy of the C5aR inhibitor CCX168 in subjects with ANCA-associated vasculitis. The aim of this trial is to test the safety and efficacy of two dose regimens of the complement C5a receptor CCX168 in patients with anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV).

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis or renal limited vasculitis
* Male and female subjects, aged at least 18 years, with new or relapsed AAV where treatment with cyclophosphamide or rituximab would be required
* Use of adequate contraception during, and for at least the three months after, any administration of study medication is required
* Positive indirect immunofluorescence (IIF) test for P-ANCA or C-ANCA, or positive ELISA test for anti-proteinase-3 (PR3) or anti-myeloperoxidase (MPO) at screening
* Have at least one "major" item, or at least 3 other items, or at least 2 renal items on the Birmingham Vasculitis Activity Score (BVAS) version 3
* Estimated glomerular filtration rate (eGFR) ≥ 20 mL per minute

Exclusion Criteria:

* Severe disease as determined by rapidly progressive glomerulonephritis, alveolar hemorrhage, hemoptysis, rapid-onset mononeuritis multiplex or central nervous system involvement
* Any other multi-system autoimmune disease
* Medical history of coagulopathy or bleeding disorder
* Received cyclophosphamide within 12 weeks prior to screening; if on azathioprine, mycophenolate mofetil, or methotrexate at the time of screening, these drugs must be withdrawn prior to receiving the cyclophosphamide or rituximab dose on Day 1
* Received intravenous corticosteroids, >3000 mg methylprednisolone equivalent, within 12 weeks prior to screening
* Received an oral daily dose of a corticosteroid of more than 10 mg prednisone-equivalent for more than 6 weeks continuously prior to the screening visit
* Received rituximab or other B-cell antibody within 52 weeks of screening or 26 weeks provided B cell reconstitution has occurred; received anti-tumor necrosis factor (TNF) treatment, abatacept, alemtuzumab, intravenous immunoglobulin (IVIg), belimumab, tocilizumab, or plasma exchange within 12 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2016-04-24 (Actual); Study Completion 2016-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (43):
- United States (39):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Long Beach, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Miami Springs, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Charlestown, Massachusetts
  - Duluth, Minnesota
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Reno, Nevada
  - Lebanon, New Hampshire
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - New Bern, North Carolina
  - Columbus, Ohio
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Canada (4):
  - Calgary, Alberta
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Lévis, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Merkel PA, Niles J, Jimenez R, Spiera RF, Rovin BH, Bomback A, Pagnoux C, Potarca A, Schall TJ, Bekker P; CLASSIC Investigators. Adjunctive Treatment With Avacopan, an Oral C5a Receptor Inhibitor, in Patients With Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. ACR Open Rheumatol. 2020 Nov;2(11):662-671. doi: 10.1002/acr2.11185. Epub 2020 Oct 31. PMID 33128347

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo BID Plus Standard of Care: Capsule, placebo, twice daily plus cyclophosphamide/rituximab plus glucocorticoids
- CCX168 10 mg BID Plus Standard of Care: Drug: CCX168 10 mg, twice daily plus cyclophosphamide/rituximab plus glucocorticoids
- CCX168 30 mg BID Plus Standard of Care: Drug: CCX168 30 mg, twice daily plus cyclophosphamide/rituximab plus glucocorticoids
Period: Overall Study
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Started | 13 | 13 | 16
Completed | 13 | 12 | 15
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care | Total
Number analyzed (Participants) | 13 | 13 | 16 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (15.42) | 60.0 (10.17) | 55.3 (13.81) | 57.7 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 9 | 23
  Male | 4 | 8 | 7 | 19
Race [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 1 | 3
  White | 13 | 11 | 14 | 38
  Other | 0 | 0 | 1 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 12 | 14 | 39
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 1 | 1 | 0 | 2
  Past smoker | 5 | 5 | 6 | 16
  Never smoked | 7 | 7 | 10 | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index
  kg/m^2 | 31.0 (12.51) | 27.6 (8.91) | 31.5 (7.59) | 30.2 (9.65)
ANCA disease status [Count of Participants; unit: Participants] — ANCA = anti-neutrophil cytoplasmic antibody ANCA status was derived from screening results that were used for subject stratification.
  Participants
    Newly diagnosed | 8 | 10 | 9 | 27
    Relapsed | 5 | 3 | 7 | 15
ANCA-associated vasculitis disease duration at screening (months) [Median (Full Range); unit: months] — If subject was relapsed, the recorded diagnosis date was used for this summary.
  months | 1.0 [0 to 95] | 1.0 [0 to 347] | 2.5 [0 to 170] | 1.0 [0 to 347]
Background treatment [Count of Participants; unit: Participants]
  Rituximab | 12 | 13 | 14 | 39
  Cyclophosphamide | 1 | 0 | 2 | 3
Type of AAV [Count of Participants; unit: Participants] — AAV = ANCA-associated vasculitis GPA = granulomatosis with polyangiitis (Wegener's)
  Participants
    GPA | 9 | 8 | 12 | 29
    Microscopic polyangiitis | 3 | 4 | 4 | 11
    Renal-limited vasculitis | 1 | 1 | 0 | 2
ANCA positivity stratification status [Count of Participants; unit: Participants] — ANCA = anti-neutrophil cytoplasmic antibody MPO = myeloperoxidase PR3 = proteinase 3
  Participants
    Anti-MPO positive | 7 | 6 | 8 | 21
    Anti-PR3 positive | 6 | 7 | 8 | 21
BVAS [Mean (Standard Deviation); unit: score on a scale] — The Birmingham Vasculitis Activity Score (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
  score on a scale | 15.0 (4.45) | 15.8 (8.84) | 15.1 (6.43) | 15.3 (6.63)
VDI score [Mean (Standard Deviation); unit: score on a scale] — The Vasculitis Damage Index (VDI) is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health)
  score on a scale | 1.2 (1.77) | 0.8 (2.49) | 0.6 (1.15) | 0.8 (1.81)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 60.1 (24.25) | 56.4 (26.75) | 61.4 (31.09) | 59.4 (27.20)
Albumin:creatinine ratio [Geometric Mean (Full Range); unit: mg/g] — Population: Only participants with values at baseline have been recorded
  mg/g
    number analyzed (Participants) | 12 | 13 | 16 | 41
    (all) | 135.4 [7 to 3262] | 76.1 [3 to 1771] | 111.9 [4 to 5540] | 104.7 [3 to 5540]
Urinary MCP-1:creatinine ratio [Geometric Mean (Full Range); unit: pg/mg creatinine] — MCP-1 = monocyte chemoattractant protein-1 Population: Only participants with values at baseline have been recorded
  pg/mg creatinine
    number analyzed (Participants) | 11 | 11 | 16 | 38
    (all) | 651.7 [162.6 to 7291.3] | 499.0 [103.3 to 3465.6] | 463.5 [97.5 to 2693.2] | 522.6 [97.5 to 7291.3]
Urinary RBCs [Count of Participants; unit: Participants] — RBC = red blood cell hpf = high power field
  Participants
    30-49 per hpf | 1 | 1 | 1 | 3
    50-75 per hpf | 1 | 1 | 0 | 2
    >75 per hpf | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: This is a safety study to assess the overall rates of treatment-emergent adverse events (TEAEs) across all study arms.
Time Frame: Baseline to Day 85
Population: Safety population: The Safety Population included all subjects who were randomized and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 13 | 16
Participants | 13 | 11 | 15

2. Primary Outcome: Proportion of Patients Achieving Disease Response Based on BVAS at Day 85
Description: Proportion of Patients achieving 50% reduction in the Birmingham Vasculitis Activity Score [BVAS] at Day 85 and no worsening in any body system component at day 85
Time Frame: Day 85
Population: ITT population: The ITT Population included all subjects who were randomized, received at least 1 dose of study medication, and had at least 1 post-baseline, on-treatment BVAS measurement.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 12 | 15
proportion of participants | 0.85 | 0.92 | 0.8

3. Secondary Outcome: Proportion of Subjects Achieving Disease Remission Based on BVAS at Day 85.
Description: Proportion of subjects achieving disease remission based on Birmingham Vasculitis Activity Score (BVAS) defined as 0 at Day 85.
Time Frame: Day 85
Population: ITT population: The ITT Population included all subjects who were randomized, received at least 1 dose of study medication, and had at least 1 postbaseline, on-treatment BVAS measurement.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 12 | 15
proportion of participants | 0.54 | 0.67 | 0.47

4. Secondary Outcome: Proportion of Subjects Achieving Early Disease Remission Based on BVAS of 0 at Days 29 and 85.
Description: Proportion of subjects achieving early disease remission based on Birmingham Vasculitis Activity Score (BVAS) score of 0 at Days 29 and 85.
Time Frame: Day 29 and 85
Population: as for outcome 3
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 12 | 15
proportion of participants | 0.15 | 0.08 | 0.2

5. Secondary Outcome: Percent Change From Baseline to Day 85 in BVAS.
Description: The Birmingham Vasculitis Activity (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health). A negative percentage change indicated improvement in health.
Time Frame: Baseline to Day 85
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 11 | 14
percentage change from baseline | -81.8 (23.30) | -95.6 (8.03) | -81.7 (31.28)

6. Secondary Outcome: Proportion of Subjects With Hematuria and Albuminuria at Baseline Who Showed a Renal Response at Day 85
Description: Renal responses among patients (who had hematuria or albuminuria at baseline determined secondary to ANCA-associated vasculitis) were defined as improvement in the following parameters of renal vasculitis: (1) increase from baseline to day 85 in eGFR [Modification of Diet in Renal Disease (MDRD equation)], (2) decrease from baseline to day 85 in hematuria (microscopic count of urinary red blood cells [RBC]), and (3) decrease from baseline to day 85 in albuminuria (first morning urinary albumin:creatinine ratio).
Time Frame: Day 85
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 6 | 5 | 8
proportion of participants | 0.17 | 0.4 | 0.63

7. Secondary Outcome: Change in Estimated Glomerular Filtration Rate at Day 85
Description: Mean Change in Estimated Glomerular Filtration Rate based on modification of diet in renal disease formula, for patients with renal disease at baseline.
Time Frame: Baseline to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 9 | 8 | 10
ml/min/1.73 m^2 | 2.0 (10.71) | 1.3 (9.75) | 6.2 (22.17)

8. Secondary Outcome: Percentage Change in Estimated Glomerular Filtration Rate at Day 85
Description: Mean Percentage Change in Estimated Glomerular Filtration Rate based on modification of diet in renal disease formula.
Time Frame: Baseline to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change from baseline (ml/min/1.73 m²)
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 9 | 8 | 10
% change from baseline (ml/min/1.73 m²) | 6.2 (35.65) | 0.9 (17.63) | 7.7 (27.92)

9. Secondary Outcome: Percent Change of Urinary Red Blood Cells in Patient With Hematuria From Baseline to Day 85
Description: Mean Percent Change of Urinary Red Blood Cells (UBC) in Patients in Hematuria at Baseline.
Time Frame: Baseline to Day 85
Population: as for outcome 2
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 7 | 5 | 8
percentage change from baseline | -56.3 [-99.67 to 100.00] | -31.5 [-99.00 to 233.33] | -95.0 [-99.38 to -81.25]

10. Secondary Outcome: Percent Change of Urinary Albumin:Creatinine Ratio in Patients With Albuminuria From Baseline to Day 85
Description: Mean Percent Change of Urinary Albumin:Creatinine Ratio in Patients with Albuminuria at Baseline
Time Frame: Baseline to Day 85
Population: as for outcome 2
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 9 | 8 | 10
percentage change from baseline | -66.281 [-92.31 to -40.40] | -13.890 [-92.86 to 175.56] | -57.596 [-96.10 to 6.03]

11. Secondary Outcome: Percent Change of Urinary MCP-1:Creatinine Ratio From Baseline to Day 85
Description: Mean Percent Change of Urinary monocyte chemoattractant protein (MCP-1:creatinine) ratio from Baseline
Time Frame: Baseline to Day 85
Population: as for outcome 2
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 11 | 9 | 14
percentage change from baseline | -33.175 [-85.20 to 106.45] | -34.802 [-87.27 to 68.48] | 63.567 [-81.63 to 1023.16]

12. Secondary Outcome: Change From Baseline to Day 85 in the VDI
Description: The Vasculitis Damage Index (VDI) is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health)
Time Frame: Baseline to Day 85
Population: ITT population: The ITT Population included all subjects who were randomized, received at least 1 dose of study medication, and had at least 1 post-baseline, on treatment BVAS measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 11 | 14
score on a scale | 0.31 (0.751) | 0.09 (0.302) | 0.14 (0.363)

13. Secondary Outcome: Change From Baseline to Day 85 in Health-Related Quality-Of-Life as Measured by the SF-36v2
Description: Change from Baseline to Day 85 in Health-Related Quality-Of-Life as Measured by the Short Form-36 (SF-36v2) SF-36v2: Medical Outcomes Survey Short Form-36 version 2. SF-36v2 measures each of the following eight health domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Scores on each item are summed and averaged. The SF-36v2 component domain scores range from 0 (worst health) to 100 (best health).
Time Frame: Baseline to Day 85
Population: ITT population: The ITT Population included all subjects who were randomized, received at least 1 dose of study medication, and had at least 1 postbaseline, on-treatment BVAS measurement.
  *p<0.05 for CCX168 compared to control for change or percent change from baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 11 | 14
score on a scale
  SF-36 Role - physical | 4.1 (11.44) | 16.1 (13.58) | 9.6 (10.15)
  SF-36 Bodily pain | -3.5 (8.40) | 11.0 (9.58) | 14.9 (7.85)
  SF-36 General health perceptions | -12.6 (4.97) | -3.8 (5.61) | -6.6 (4.49)
  SF-36 Vitality | -2.5 (8.09) | 13.8 (9.31) | 11.8 (7.38)
  SF-36 Social functioning | 4.4 (7.81) | 15.2 (8.96) | 0.5 (7.12)
  SF-36 Mental health | 8.2 (5.49) | 13.3 (5.80) | 12.6 (4.66)
  SF-36 Reported health transition | -0.7 (0.48) | -1.1 (0.58) | -1.6 (0.44)
  SF-36 Physical functioning | 4.9 (7.51) | 13.5 (8.33) | 17.2 (6.61)
  SF-36 Role - emotional | 8.4 (7.76) | 10.8 (8.42) | 12.7 (6.80)

14. Secondary Outcome: Mean Change From Baseline to Day 85 in Health-related Quality-of-life as Measured by the EQ-5D-5L
Description: Mean Change from baseline to Day 85 in health-related quality-of-life as measured by the Euro Quality-of-Life-5 Domains-5 Levels (EQ-5D-5L).
  EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given can be converted into an Index Score ranging from 0 for death to 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Baseline to Day 85
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 11 | 14
score on scale
  EQ-5D-5L VAS Score | 12.85 (25.413) | 20.18 (18.121) | 11.21 (21.641)
  EQ-5D-5L Index Score | 0.03 (0.140) | 0.05 (0.200) | 0.04 (0.138)

15. Secondary Outcome: Proportion of Subjects Requiring Rescue Glucocorticoid Treatment From Baseline to Day 85
Description: Proportion of subjects requiring rescue glucocorticoid treatment from Baseline to Day 85
Time Frame: Baseline to Day 85
Population: as for outcome 3
Measure: Number; unit: proportion of participants
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
Number analyzed (Participants) | 13 | 13 | 16
proportion of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to day 169
Description: The Safety Population included all subjects who were randomized and received at least 1 dose of study drug
Arm/Group | Placebo BID Plus Standard of Care | CCX168 10 mg BID Plus Standard of Care | CCX168 30 mg BID Plus Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/13 | 2/13 | 4/16
Other Adverse Events (participants affected / at risk) | 13/13 | 12/13 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID Plus Standard of Care (N=13) | CCX168 10 mg BID Plus Standard of Care (N=13) | CCX168 30 mg BID Plus Standard of Care (N=16)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (General disorders) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID Plus Standard of Care (N=13) | CCX168 10 mg BID Plus Standard of Care (N=13) | CCX168 30 mg BID Plus Standard of Care (N=16)
Oedema peripheral (General disorders) | 1 | 2 | 4
Fatigue (General disorders) | 3 | 2 | 1
Pain (General disorders) | 0 | 1 | 1
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 4 | 3 | 4
Hot flush (Vascular disorders) | 0 | 1 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2
Amylase increased (Investigations) | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 1 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Scleritis (Eye disorders) | 0 | 1 | 1
Conjunctival hemorrhage (Eye disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Thirst (General disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0
Dystonia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1
Blood bicarbonate increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study had a small sample size and was not powered to detect differences between avacopan or placebo arms or among subgroups of patients such as newly-diagnosed vs. relapsed status, or on the basis of characteristics such as ANCA type.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02222155/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02222155/SAP_001.pdf